CLINICAL TRIAL: NCT04914026
Title: MicroRNA-371 as Markers for Disease Activity and as a Tool to Monitor the Effect of Chemotherapy and Early Detection of Recurrence in Patients With Testicular Germ Cell Tumours
Brief Title: MicroRNA as Markers in Testicular Cancer
Status: Recruiting | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Collaborators: Karolinska University Hospital (Other); Sahlgrenska University Hospital (Other); Helse Fonna (Other); University Hospital of North Norway (Other); Oslo University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2015/1475
Record Dates: First submitted 2021-05-31; First posted 2021-06-04 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Testicular Germ Cell Cancer; Seminoma; Non-Seminoma Testicular Cancer; Stage I Testicular Cancer; Stage II Testicular Cancer; Stage III Testicular Cancer; Stage IV Testicular Cancer; Relapse Testicular Cancer
MeSH Terms: conditions — Testicular Neoplasms; Seminoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood is collected in order to extract RNA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Biomarker analysis — Blood collection. Blood samples will be collected at diagnosis, during surveillance, during treatment and every 3-6 months

SUMMARY:
The main objective of this study is establish the performance of miR371 in management of testicular cancer

DETAILED DESCRIPTION:
The main objective of the study is to asses the sensitivity and specificity of microRNA-371a-5p (miR371) in detection of viable testicular germ tumour cells. To assess the utility of miR371 at orchiectomy, during treatment and surveillance and in early detection of recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected testicular cancer, referred to orchiectomy.
* Patients diagnosed with testicular germ cell cancer.
* Age 18-70 years of age.
* Must be able receive information and to consent.

Exclusion Criteria:

* Other prior or concomitant malignancy (other than testicular cancer).
* Other diseases or conditions that hinder the ability to receive information and to participate in follow-up procedures.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Testicular Germ Cell Cancer
Study Population: Men with suspected and confirmed testicular germ cell cancer, aged 18-70 years. Seminomas and non-seminomas, stage I-IV.
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2016-12-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
miR371 as a biomarker in testicular germ cell cancer at orchiectomy | 5 years
  To estimate the sensitivity and specificity of miR371 in identifying viable tumour cells at diagnosis
miR371 as a biomarker in testicular germ cell cancer at RPLND | 5 years
  To estimate the sensitivity and specificity of miR371 in identifying viable tumour cells at RPLND
miR371 as a biomarker in testicular germ cell cancer during chemotherapy treatment | 5 years
  To estimate the performance of miR371 in monitoring of treatment efficiency (chemotherapy)
miR371 as a biomarker in testicular germ cell cancer and detection of recurrence | 5 years
  To estimate the performance of miR371 in (early) detection of recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Mette Pernille Myklebust, PhD, Principal Investigator — Haukeland University Hospital
Locations (6):
- Norway (4):
  - Haukeland University Hospital, Bergen
  - Haugesund Hospital, Haugesund
  - Oslo University Hospital, Oslo
  - University Hospital of North Norway, Tromsø
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Karolinska University Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: No